CLINICAL TRIAL: NCT07146386
Title: A Randomized, Double-blind, Controlled, Non-inferiority Multicenter Phase III Clinical Study Evaluating the Efficacy and Safety of H077 Sustained-release Tablets Versus Silodosin Capsules in the Treatment of Benign Prostatic Hyperplasia
Brief Title: A Phase III Clinical Study of H077 Sustained-Release Tablets Compared With Silodosin Capsules in the Treatment of Benign Prostatic Hyperplasia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Huilun Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-H077-III-01
Record Dates: First submitted 2025-08-12; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostatic Hyperplasia; Benign Prostatic Hyperplasia With Lower Urinary Tract Symptoms
Keywords: Benign prostatic hyperplasia; lower urinary tract symptoms; Silodosin; selective α1A-adrenergic receptor blocker; IPSS scores
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — silodosin; Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, randomized, double-blind, controlled non-inferiority phase III study, evaluating the efficacy and safety of H077 sustained-release tablets compared with silodosin capsules in the treatment of benign prostatic hyperplasia (BPH).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- H077 treatment group (Experimental): Subjects are administered one H077 sustained-release tablet (8 mg) orally once daily, along with one silodosin capsule (placebo) orally twice daily.
  Interventions: Drug: H077 sustained-release tablet
- Silodosin capsules Control Group (Active Comparator): Subjects are administered one Silodosin capsule (4 mg) twice daily, along with one H077 sustained-release tablet placebo once daily, orally.
  Interventions: Drug: Silodosin capsules Control Group

INTERVENTIONS:
Drug: H077 sustained-release tablet — Subjects are administered one H077 sustained-release tablet (8 mg) orally once daily, along with one silodosin capsule (placebo) orally twice daily.
  Arms: H077 treatment group
Drug: Silodosin capsules Control Group — Subjects are administered one Silodosin capsule (4 mg) twice daily, along with one H077 sustained-release tablet placebo once daily, orally.
  Arms: Silodosin capsules Control Group

SUMMARY:
This is a randomized, double-blind, controlled, non-inferiority multicenter Phase III clinical study to evaluate the efficacy and safety of H077 sustained-release tablets versus silodosin capsules in treating benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 50 to 75 years old, inclusive of both endpoints;
2. Meets the clinical diagnostic criteria for benign prostatic hyperplasia (BPH);
3. IPSS score was ≥ 8 points, and the QOL score was ≥ 3 points during the screening period;
4. Prostate volume ≥ 20 ml (measured by transabdominal ultrasound);
5. PSA≤4 ng/mL;
6. During the screening period, Qmax > 5 ml/s and Qmax <15 ml/s (urine output ≥ 125 ml);
7. The subjects had no intention of having children from the screening stage until 6 months after the last administration of the drug, and they were able to take effective contraceptive measures;
8. Understand and voluntarily sign the written informed consent form (ICF), and be willing and capable of undergoing regular visits, treatment plans, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Those who are allergic to any component of α/β-adrenergic receptor blockers or the test drugs; or who have contraindications;
2. History or evidence of prostate cancer (such as positive biopsy or ultrasound result, suspicious DRE findings), excluding patients who had suspicious ultrasound or DRE findings within 6 months prior to the screening but had negative biopsy results and stable PSA levels;
3. During the screening process, researchers identified patients with BPH who required minimally invasive prostate treatment or surgical intervention;
4. Has previously undergone prostate surgery, including open prostate surgery, transurethral minimally invasive prostate surgery, balloon dilation or stent replacement, or other invasive measures for treating BPH;
5. Subjects with residual urine volume greater than 100 mL (measured by transabdominal ultrasound) or those for whom catheterization is deemed necessary by the investigator;
6. Subjects who underwent cystoscopy, other transurethral endoscopic procedures, or therapeutic urinary catheterization within 1 month prior to the screening period;
7. Subjects with a history of acute urinary retention (AUR) or cystostomy within 3 months prior to the screening period;
8. Subjects with documented pelvic cavity trauma or urethral surgical interventions;
9. During the screening period, any disease other than BPH that the investigator deems could cause urinary symptoms or changes in urine flow rate (such as neurogenic bladder, bladder neck fibrosis, bladder tumor, urinary calculi, urethral stricture, phimosis or penile tumor, acute or chronic prostatitis, acute or chronic urinary tract infection, acute or chronic renal failure, congenital developmental abnormalities of the urinary and reproductive system, etc.) must be excluded;
10. During the screening period, subjects with positive hepatitis B surface antigen (HBsAg) and HBV-DNA levels greater than 500 IU/ml, or with positive hepatitis C virus antibody (HCV-Ab) and HCV-RNA levels greater than 500 IU/ml, or who had received hepatitis-related antiviral drug treatment within 6 months prior to the first administration;
11. During screening period, the levels of aspartate transaminase (AST) or alanine transaminase (ALT) were more than 3 times the upper limit of the normal range;
12. During the screening period, serum creatinine was greater than 1.5 times the upper limit of the normal range;
13. Patients who plan to undergo cataract surgery during the medication period and within 3 months after the medication is completed;
14. Currently or previously have the following diseases or conditions: a) Have a clear history of orthostatic hypotension in the past, or have a positive orthostatic hypotension test; or have a history of malignant hypertension; b) Have recurrent dizziness, vertigo, loss of consciousness or syncope, or any other signs or symptoms that the investigator considers may be worsened by celerodisonic; c) Have undergone major surgery (excluding biopsy) within 4 weeks before screening and have not fully recovered; d) Have had myocardial infarction, unstable angina pectoris, need for clinical intervention or clinical symptoms of arrhythmia, need for clinical intervention or clinical symptoms of congestive heart failure, or any cerebrovascular accident within 6 months before screening; e) Have a previous surgical history or have severe gastrointestinal diseases, which the investigator considers may affect the absorption, distribution, metabolism, etc. of the study drug; f) Have active infectious diseases and require systemic anti-infection treatment; g) Have a history of diabetes and poor blood sugar control, or have patients with diabetic nephropathy that require drug control; h) Have had malignant tumors within 5 years before screening; i) Have patients with other serious primary diseases and functional disorders in the heart, brain, lungs, liver, kidneys, hematopoietic system, endocrine system, etc;
15. Currently or previously used the following drugs: a) Within 3 months before screening or during the study, need to use 5α-reductase inhibitors, anti-androgen drugs, and androgen drugs or any other drugs that affect hormone levels or prostate volume; b) Within 2 weeks before screening or during the study, need to use any α-adrenergic receptor blockers or any α-receptor blockers other than cilorodin during the study; c) Within 4 weeks before screening or during the study, need to use PDE-5 inhibitors, anticholinergic drugs, anticholinergic drugs or any other drugs that affect urinary function; d) Within 2 weeks before screening or during the study, need to use traditional Chinese medicine, Chinese herbs, or botanical preparations with indications for BPH; e) Within 4 weeks before screening or during the study, need to use any CYP3A4 strong inhibitors, CYP3A4 strong inducers or P-gp strong inhibitors;
16. Subjects who participated in other drug or device clinical trials within 3 months prior to screening;
17. Subjects with current alcohol or substance abuse were excluded;
18. The researchers determined that the patient had other circumstances that affected the safety or efficacy assessment of the study drug, the obtaining of informed consent, or the compliance with the study procedures.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 728 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
changes in International Prostatism Symptom Score (IPSS) at 12 weeks from baseline | baseline to 12 weeks
  The study set the change in the IPSS of patients after 12 weeks of medication compared to the baseline data as the primary endpoint. The IPSS is currently the internationally recognized best method for assessing the severity of symptoms in patients with benign prostatic hyperplasia. The IPSS scale is used to evaluate the severity of 7 urinary symptoms, namely: incomplete urination, frequent urination, intermittent urine flow, urgency, weak urine stream, difficulty in urination, and nocturia frequency. Each of the 7 symptoms is scored in 6 segments based on the occurrence in the last month (0-5 points, 0 indicates no occurrence, 5 indicates almost always occurring). The total score is 35 points, and the patient's symptoms are classified as mild (0-7 points), moderate (8-19 points), and severe (20-35 points).

SECONDARY OUTCOMES:
changes in IPSS at 1, 2, 4, and 8 weeks from baseline | baseline to 1, 2, 4, and 8 weeks
  The changes in the IPSS compared to the baseline after 1, 2, 4, and 8 weeks of medication administration.
quality of life (QOL) scores | baseline to 1, 2, 4, 8, and 12 weeks
  The QOL score is used to understand the patient's subjective perception of their current level of lower urinary tract symptoms throughout their lifetime. It mainly focuses on the extent to which BPH patients are troubled by lower urinary tract symptoms and whether they can tolerate it. Based on subjective feelings, it is classified as: happy, satisfied, generally satisfied, acceptable, not very satisfied, distressed, and very bad. The scores range from 0 to 6.
The proportion of subjects whose IPSS scores changed by ≥ 3 points or improved by ≥ 25% compared to the baseline | baseline to 1, 2, 4, 8, and 12 weeks
  The proportion of subjects whose IPSS scores changed by ≥ 3 points or improved by ≥ 25% compared to the baseline after 1, 2, 4, 8, and 12 weeks of medication administration.
maximum urine flow rate (Qmax) changes | baseline to 2, 4, 8, and 12 weeks
  The changes in the maximum urine flow rate (Qmax) compared to the baseline after 2, 4, 8, and 12 weeks of medication administration.
The proportion of subjects whose Qmax increased by ≥ 3 ml/s and improved by ≥ 30% compared to the baseline | baseline to 1, 2, 4, 8, and 12 weeks
  The proportion of subjects whose Qmax increased by ≥ 3 ml/s and improved by ≥ 30% compared to the baseline after 1, 2, 4, 8, and 12 weeks of medication administration.
The incidence of acute urinary retention (AUR) during medication administration | baseline to 12 weeks
  The incidence of acute urinary retention (AUR) during medication administration
The incidence of BPH-related surgical treatment. | baseline to 12 weeks
  The proportion of participants who discontinued the study treatment during the medication period due to the need for BPH-related surgical treatment.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | baseline to 13 weeks
  the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), as well as changes in vital signs and laboratory test results, etc.
Multiple-dose exposure-response relationship | baseline to 1, 2, 4, 8, and 12 weeks
  Trough plasma concentrations will be measured after multiple oral doses of H077 sustained-release tablets in BPH subjects. Individual systemic exposure will be predicted from trough concentrations and subsequently utilized for exposure-response analysis.

CONTACTS AND LOCATIONS:
Locations (66):
- China (66):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial People's Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - The Tenth Affiliated Hospital of Southern Medical University (Dongguan People's Hospital), Dongguan, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - First Affiliated Hospital of Hebei University of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - The People's Hospital of Anyang City, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The Sixth hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Wuhan Hospital of Traditional Chinese And Western Medicine, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital affiliated to Nanjing Medical University, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - Affiliated Hospital of Jiujiang University, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Jining First People's Hospital, Jining, Shandong
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - Chengdu Xindu District People's Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Third People's Hospital of Chengdu, Affiliated Hospital of Southwest Jiaotong University, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang Uygur Autonomous Region
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Huzhou First People's Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - The Fourth Hospital of Zhejiang University School of Medicine, Jinhua, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No